CLINICAL TRIAL: NCT06629948
Title: Correlation Between the Cobb's Angle and the Forward Head Posture in Patients With Adolescent Idiopathic Scoliosis
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Ezzat Ibrahim Aziz, DR, Cairo University
Other Study IDs: Forward head in AIS
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS); Forward Head Posture
Keywords: Forward head; scoliosis; craniovertebral angle
MeSH Terms: conditions — Scoliosis | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: x ray — whole spine x ray posterioanterior and lateral views
Diagnostic Test: the cranio-cervical flexion test — measure of deep neck flexors muscles endurance

SUMMARY:
Purpose of This study to detect if there is correlation between the Cobb's angle and the forward head posture in patients with Adolescent Idiopathic Scoliosis.

And if there is correlation between the Cobb's angle and the cervical sagittal curve angle in AIS. And also if there is correlation between the Cobb's angle and deep flexors muscles endurance in AIS

DETAILED DESCRIPTION:
The prevalence of sagittal profile imbalance in adolescent idiopathic scoliosis is not known exactly as little research is available in this context (Nasser et al., 2023) Thought based on previous studies that a forward head corrective exercise program combined with conventional rehabilitation improved three-dimensional scoliotic posture and functional status in patients with adolescent idiopathic scoliosis. (Alia Diab et al., 2012) Up to our knowledge there is no significant evidence that there is correlation between Craniovertebral angle (CVA) and idiopathic scoliosis by Cobb's angle.

So we need to make a simple assessment method of the severity of scoliosis and its impact on head position through a simpler method by observing the cervical curvature through photos for CVA, This can help to avoid unnecessary radiological examination. In addition, it also may help in paying the attention to the correction of cervical spines, head position and cervical muscles endurance during conservative treatment of scoliosis.

Also studying cervical sagittal alignment deformities will help in surgical operations to maintain or restore sagittal physiological curvature side by side with correction of coronal scoliosis angle in order to prevent adjacent segment degeneration after the fusion operation.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patients with AIS. 2- Patient with forward head posture CVA less than 48 degress. (Fard et al .,2021) 3- Patients aged between 10 and 18 years, (Upasani et al., 2007). 4- Patients who underwent Posterioanterior (PA) and lateral X-ray radiography, and Cobb angle >10°.(Nasser et al.,2023) 5- Patients with Lenke types (1 to 6). 6- No previous spine surgery ((Wang, et al., 2017).

Exclusion Criteria:

* 1- Patients with congenital scoliosis (including hemivertebrae, butterfly vertebrae, and failure of segmentation), (Shu-Man Han et al., 2022 and Nasser et al., 2023).

  2- Other developmental thoracic deformity (funnel chest etc.). 3- Scoliosis with definitive reasons (secondary to neurofibromatosis, Marfan syndrome, and syringomyelia).

  4- Patients with neurologic deficit or spondylolisthesis (Upasani et al., 2007).

  5- History of spinal trauma and infection, and metabolic bone disease.

Ages: 10 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Thirty four Male and female subjects with adolescent idiopathic scoliosis participating in this study will be assigned homogenously some of them with Cobb's angle below 45 degrees and others above 45 degrees (n=34) and they will sign a consent form.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
1- Measurement of Craniovertebral angle CVA | within 3 months from enrollment
  We will measure The Craniovertebral angle by the photogrammetric method
Measurement of Cobb's angle | within 3 months from enrollment
  Measurement of Cobb's angle from whole spine xray
Measurement of sagittal cervical curve angle | within 3 months from enrollment
  Measurement of cervical spines sagittal curve from lateral view X-ray
4- Measurement of deep flexors muscle endurance. | within 3 months from enrollment
  Activation and performance scores will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy Youssef, Professor, Principal Investigator — Professor and chairperson of Department of Orthopaedic Physical Therapy for Musculoskeletal Disorders and its Surgery Faculty of Physical Therapy Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yaman O, Dalbayrak S. Idiopathic scoliosis. Turk Neurosurg. 2014;24(5):646-57. doi: 10.5137/1019-5149.JTN.8838-13.0. PMID 25269032
- [Background] Latalski M, Danielewicz-Bromberek A, Fatyga M, Latalska M, Krober M, Zwolak P. Current insights into the aetiology of adolescent idiopathic scoliosis. Arch Orthop Trauma Surg. 2017 Oct;137(10):1327-1333. doi: 10.1007/s00402-017-2756-1. Epub 2017 Jul 14. PMID 28710669
- [Background] Yip CH, Chiu TT, Poon AT. The relationship between head posture and severity and disability of patients with neck pain. Man Ther. 2008 May;13(2):148-54. doi: 10.1016/j.math.2006.11.002. Epub 2007 Mar 23. PMID 17368075
- [Background] Wang L, Liu X. Cervical sagittal alignment in adolescent idiopathic scoliosis patients (Lenke type 1-6). J Orthop Sci. 2017 Mar;22(2):254-259. doi: 10.1016/j.jos.2016.12.006. Epub 2016 Dec 23. PMID 28025024
- See also: Related Info — https://journals.lww.com/spinejournal/fulltext/2007/05200/analysis_of_sagittal_alignment_in_thoracic_and.16.aspx